CLINICAL TRIAL: NCT04306562
Title: Effect of Oral Protein Supplementation on Postoperative Complications in Elderly Sarcopenic Cancerous Patients: A Randomized Controlled Trial
Brief Title: Effect of Oral Protein Supplementation on Postoperative Complications in Elderly Sarcopenic Cancerous Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The clinical study was terminated prior to completion due to challenges in enrolling a sufficient number of participants.
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Associated Professor, Siriraj Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB632
Record Dates: First submitted 2020-03-09; First posted 2020-03-13 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Sarcopenia; Cancer
Keywords: Protein supplementation; Perioperative
MeSH Terms: conditions — Sarcopenia; Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients who were diagnosed with sarcopenia or severe sarcopenia, will be randomly assigned following stratified randomization procedures (computerized random numbers) to one of two groups.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The allocation sequence will be concealed from the researcher enrolling and assessing participants in sequentially numbered, opaque, sealed and stapled envelopes. Corresponding envelopes will be opened only after the enrolled participants completed all baseline assessments and it was time to allocate the intervention. Whereas patients and physicians allocated to the intervention group are aware of the allocated arm, outcome assessors and data analysts will be kept blinded to the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients in an intervention group will be ask about a history of food consumption in the past seven days to analyze a nutritive value of food consumption with a program (INMUCAL-Nutrients V.4.0, Institute of Nutrition, Mahidol University) and estimate an enteral nutrition supplement to reach a target of total dietary protein intake of 1.5 g/kg/day with nutritional counseling by researchers. Special enteral formula will be selected if patients have specific conditions including renal failure, hyperglycemia/diabetes and liver failure, acute and chronic pulmonary disease and immunocompromised states. Otherwise, standard formula will be provided. Duration of enteral protein supplementation is at least 14 days from a preanesthetic clinic visit to a day of surgery.
  Interventions: Dietary Supplement: enteral nutrition supplement
- Control group (No Intervention): Patients in a control group will be sent to assess and improve nutritional status by primary doctor as a conventional care pathway.

INTERVENTIONS:
Dietary Supplement: enteral nutrition supplement — enteral nutrition supplement to reach a target of total dietary protein intake of 1.5 g/kg/day for at least 14 days from a preanesthetic clinic visit to a day of surgery.
  Arms: Intervention group

SUMMARY:
Sarcopenia is a condition of reduced skeletal muscle associated with aging. It leads to poor outcome and increased risk of postoperative complications. Achieving protein and energy requirements is crucial point in sarcopenia treatment. In preoperative patients, daily consumption of protein should be at least 1.2-2.0 g of protein/kg/day or 25-35 g of protein in a meal to provide muscular protein synthesis.

The objective of this study is to show that preoperative enteral protein supplementation in elderly cancerous patients, who are diagnosed with sarcopenia, can decrease morbidity such as postoperative complications; mortality and improve postoperative clinical outcomes after elective surgery.

DETAILED DESCRIPTION:
Sarcopenia is a condition of reduced skeletal muscle mass associated with aging process leading to decrease muscle strength and function. International Working Group on Sarcopenia defines Sarcopenia as an age-associated loss of skeletal muscle mass and function, and the European Working Group on Sarcopenia in Older People (EWGSOP) defines sarcopenia as a syndrome characterized by progressive and generalized loss of skeletal muscle mass and strength with a risk of adverse outcomes such as physical disability, poor quality of life, and death. The prevalence of sarcopenia is higher in population older than 65 years and leading to poor outcomes such as mobility disorders, disability, poor quality of life and death. Sarcopenia is also associated with an increased risk of postoperative complications such as overgrowth of bacteria in the gastrointestinal tract, postoperative infections, sepsis, delayed wound healing prolonged inpatient rehabilitation, mortality and consequently a longer length of hospital stay, even without nutritional risk.

Sarcopenia contains multifactorial etiology, such as age-related, inadequate energy and/or protein intake, sedentary activity such as bed rest, and coexisting disease such as organ failure, inflammatory disease or endocrine disease. One important goal of developing treatment strategies in sarcopenic patients is to achieve protein and energy requirements. In preoperative patients, daily consumption of protein should be at least 1.2-2.0 g of protein/kg/day or 25-35 g of protein in a meal to provide muscular protein synthesis. Perioperative oral protein supplements have been demonstrated to increase serum albumin and total protein, improve postoperative functional walking capacity and decrease postoperative infection in elderly or critically ill patients. However, there have been no studies on the benefit of preoperative protein supplement in cancerous patients.

The objective of this study is to show that preoperative enteral protein supplementation in elderly cancerous patients, who are diagnosed with sarcopenia, can decrease morbidity such as postoperative complications; mortality and improve postoperative clinical outcomes after elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age of equal or more than 65 years.
* Diagnosed cancer of gastrointestinal tract, hepatopancreaticobiliary tract, urology, head and neck, ear-nose-throat or gynecological cancer.
* Scheduled for elective surgery with the duration more than 2 hours will be enrolled in this study.

Exclusion Criteria:

* Unable to walk, stand up, perform hand grip test, communicate and follow commands.
* Having factors affect bioimpedance (BIA) analysis such as pacemaker, alcohol drinking or heavy exercise within 12 hours prior to analysis or take medication, herb or hormone that affect muscle mass and strength such as estrogen, testosterone, thyroxine, steroid.
* Patients diagnosed with no sarcopenia or probable sarcopenia or have a contraindication for enteral nutrition will be excluded from this study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | 30 days after operation
  postoperative complications within 30 days after operation which will be recorded and classify into surgical or non-surgical complications. All complication will be graded using Dindo-Clavien classification into 5 grades; Grade I is any deviation from the normal postoperative course without the need for pharmacological treatment or surgical, endoscopic, and radiological interventions; Grade II is complication which requiring pharmacological treatment with drugs (other than such allowed for grade I), blood transfusions or total parenteral nutrition are also included; Grade III requires surgical, endoscopic or radiological intervention; Grade IV is life-threatening complication (including CNS complications) requiring ICU management; Grade V means death of a patient.

SECONDARY OUTCOMES:
mortality rate | 90 days after operation
  number of patient death within 90 days after operation of elective surgery
duration of hospital admission | through patients discharge, an average of 1 week
  duration of hospital admission record in days.

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fielding RA, Vellas B, Evans WJ, Bhasin S, Morley JE, Newman AB, Abellan van Kan G, Andrieu S, Bauer J, Breuille D, Cederholm T, Chandler J, De Meynard C, Donini L, Harris T, Kannt A, Keime Guibert F, Onder G, Papanicolaou D, Rolland Y, Rooks D, Sieber C, Souhami E, Verlaan S, Zamboni M. Sarcopenia: an undiagnosed condition in older adults. Current consensus definition: prevalence, etiology, and consequences. International working group on sarcopenia. J Am Med Dir Assoc. 2011 May;12(4):249-56. doi: 10.1016/j.jamda.2011.01.003. Epub 2011 Mar 4. PMID 21527165
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Background] Cruz-Jentoft AJ, Landi F, Topinkova E, Michel JP. Understanding sarcopenia as a geriatric syndrome. Curr Opin Clin Nutr Metab Care. 2010 Jan;13(1):1-7. doi: 10.1097/MCO.0b013e328333c1c1. PMID 19915458
- [Background] Chen LK, Liu LK, Woo J, Assantachai P, Auyeung TW, Bahyah KS, Chou MY, Chen LY, Hsu PS, Krairit O, Lee JS, Lee WJ, Lee Y, Liang CK, Limpawattana P, Lin CS, Peng LN, Satake S, Suzuki T, Won CW, Wu CH, Wu SN, Zhang T, Zeng P, Akishita M, Arai H. Sarcopenia in Asia: consensus report of the Asian Working Group for Sarcopenia. J Am Med Dir Assoc. 2014 Feb;15(2):95-101. doi: 10.1016/j.jamda.2013.11.025. PMID 24461239
- [Background] Simonsen C, de Heer P, Bjerre ED, Suetta C, Hojman P, Pedersen BK, Svendsen LB, Christensen JF. Sarcopenia and Postoperative Complication Risk in Gastrointestinal Surgical Oncology: A Meta-analysis. Ann Surg. 2018 Jul;268(1):58-69. doi: 10.1097/SLA.0000000000002679. PMID 29373365
- [Background] Reisinger KW, van Vugt JL, Tegels JJ, Snijders C, Hulsewe KW, Hoofwijk AG, Stoot JH, Von Meyenfeldt MF, Beets GL, Derikx JP, Poeze M. Functional compromise reflected by sarcopenia, frailty, and nutritional depletion predicts adverse postoperative outcome after colorectal cancer surgery. Ann Surg. 2015 Feb;261(2):345-52. doi: 10.1097/SLA.0000000000000628. PMID 24651133
- [Background] Kuwada K, Kuroda S, Kikuchi S, Yoshida R, Nishizaki M, Kagawa S, Fujiwara T. Sarcopenia and Comorbidity in Gastric Cancer Surgery as a Useful Combined Factor to Predict Eventual Death from Other Causes. Ann Surg Oncol. 2018 May;25(5):1160-1166. doi: 10.1245/s10434-018-6354-4. Epub 2018 Feb 5. PMID 29404820
- [Background] Friedman J, Lussiez A, Sullivan J, Wang S, Englesbe M. Implications of sarcopenia in major surgery. Nutr Clin Pract. 2015 Apr;30(2):175-9. doi: 10.1177/0884533615569888. Epub 2015 Feb 13. PMID 25681482
- [Background] Ma BW, Chen XY, Fan SD, Zhang FM, Huang DD, Li B, Shen X, Zhuang CL, Yu Z. Impact of sarcopenia on clinical outcomes after radical gastrectomy for patients without nutritional risk. Nutrition. 2019 May;61:61-66. doi: 10.1016/j.nut.2018.10.025. Epub 2018 Oct 24. PMID 30703570
- [Background] Lieffers JR, Bathe OF, Fassbender K, Winget M, Baracos VE. Sarcopenia is associated with postoperative infection and delayed recovery from colorectal cancer resection surgery. Br J Cancer. 2012 Sep 4;107(6):931-6. doi: 10.1038/bjc.2012.350. Epub 2012 Aug 7. PMID 22871883